CLINICAL TRIAL: NCT02286791
Title: Mindful Awareness Program for the Prevention of Dementia: A Randomized Controlled Trial
Acronym: MAPRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Rathi Mahendran, Senior Consultant Psychiatrist, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B-14-110
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Dementia
Keywords: Prevention of dementia; Mindful awareness program; Mild cognitive impairment; Mindfulness; Elderly; Cognitive decline
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindful Awareness Program (Experimental): 18 sessions of mindful awareness program teaching the elderly mindful awareness practice techniques
  Interventions: Behavioral: Mindful Awareness Program
- Health Education Program (Active Comparator): 18 sessions of health education program focusing on healthy living topics
  Interventions: Behavioral: Health Education Program

INTERVENTIONS:
Behavioral: Mindful Awareness Program — For Mindful Awareness Program, 40-minutes weekly sessions for 12 weeks, followed by 40-minutes monthly for 6 months. The mindful awareness practice techniques to be taught to the elderly include: (1) mindfulness of the senses practice; (2) the body scan practice; (3) walking meditation practice; (4) 'movement nature meant' practice; and (5) visuo-motor limb tasks
  Other Names: MAP
  Arms: Mindful Awareness Program
Behavioral: Health Education Program — For the Health Education Program, weekly sessions of 40 minutes for 12 weeks, followed by monthly sessions of 40 minutes for 6 months.
  Week 1: Diabetes Mellitus Week 2: Hypertension Week 3: Home Safety Week 4: Medications Week 5: Diet Week 6: Depression Week 7: Dementia Week 8: Anxiety Week 9: Sleep Week 10: Exercise Week 11: Coping with bereavement Week 12: Social support
  Other Names: HEP
  Arms: Health Education Program

SUMMARY:
The objective of this study is to determine whether regular Mindful Awareness Program (MAP) may reverse cognitive impairment and/or prevent further cognitive decline among older adults. 60 elderly with mild cognitive impairment (MCI) were randomized to participate in either the MAP or the Health Education Program (HEP). Sessions will be conducted weekly for 12 weeks, and monthly for 6 months. Participants would be assessed at 3 time-points: at the start, at 3-months and at 9-months.

It was hypothesized that as compared to HEP participants, MAP participants will (1) have improved functional connectivity, (2) have a decreased risk in cognitive decline and (3) report higher psychological well-being.

DETAILED DESCRIPTION:
Participants Study participants are community-dwelling elderly.

Assessments Demographic data will be collected at the start. Psychological tests for depression and anxiety and neuropsychological tests of cognitive functioning will be done at the start, at 3-months and at 9-months, the end of the study. A urine sample will be collected at the start and at the end of the study; blood, fecal and saliva samples will be collected at all three time points. Participants will also undergo a brain neuro-imaging scan at the start of the study and at the 3-months interval.

Intervention Sessions This is an intervention study with a control group design. The strength of this design is its experimental nature with randomization. The control group is the health education program participants.

In the Mindful Awareness Program, all 30 participants will be seen in a group format once a week for 40 minutes for 12 weeks, followed by once a month for 40 minutes for 6 months. The intervention is modelled on similar groups teaching mindfulness meditation to the elderly. The sessions will be led by an experienced instructor who has conducted pilot studies on the use of mindful awareness practice techniques with the elderly.

Participants shall be required to practice these techniques at home daily and will be asked to keep a log of their practice.

For the Health Education Program, all 30 participants will be seen in a group format once a week for 40 minutes for 12 weeks, followed by once a month for 40 minutes for 6 months. Each weekly session will cover a healthy living topic related to maintaining and improving cognitive function. The monthly sessions will review the topics covered with a discussion of how participants have implemented the imparted knowledge to their daily lives. The sessions will be led by an experienced instructor who has conducted similar teaching sessions to the elderly.

Participants will be provided with hand-outs at each session, and there will be discussions to encourage them to practice what is being taught in their daily lives.

ELIGIBILITY:
Inclusion Criteria:

1. an elderly person between the age of 60 and 85 living in the community and fulfill the operational criteria/definition of MCI:

   1. At least one age-education adjusted neuropsychological test Z score < -1.5
   2. Do not meet DSM-IV criteria for dementia syndrome
   3. Memory / Cognitive complaint, preferably corroborated by a reliable informant
   4. Intact Activities of Daily Living.
2. function independently
3. do not suffer from dementia,
4. able to travel on their own to the data collection site and participate in the MAP or HEP

Exclusion Criteria:

1. Those who do not meet the above inclusion criteria (ie. Do not have a MCI diagnosis),
2. Those with Dementia or Normal Ageing
3. Have a neurological condition (e.g., epilepsy, Parkinson's Disease),
4. Have a major psychiatric condition (e.g., major depressive disorder)
5. Suffer from a terminal illness (e.g., cancer).
6. Have significant visual or hearing impairment, or
7. Marked upper and lower limb motor difficulties, which may affect their ability to participate in the study.
8. Are in another interventional study at the same time

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline Mini-Mental State Examination (MMSE) at 3 months and 9 months | baseline, 3-months, 9-months
  Mini-Mental State Examination (MMSE) is a brief 30-point questionnaire administered by health care professionals to screen for cognitive impairment. The score ranges from 0 to 30; the higher the score, the less impaired is the participant's cognitive function.
Change from baseline Clinical Dementia Rating (CDR ) at 3 months and 9 months | baseline, 3-months, 9-months
  Clinical Dementia Rating (CDR ) is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias: Memory, Orientation, Judgment & Problem Solving, Community Affairs, Home & Hobbies, and Personal Care.
Change from baseline Rey Auditory Verbal Learning Test (RAVLT) at 3 months and 9 months | baseline, 3-months, 9-months
  Rey Auditory Verbal Learning Test (RAVLT) evaluates declarative verbal learning and memory.
Change from baseline Digit Span Task at 3 months and 9 months | baseline, 3-months, 9-months
  Digit Span Task, which consists of a Digit Span Forward (DSF) and a Digit Span Backward (DSB) task is used to assess attention and verbal working memory.
Change from baseline Colour Trails Tests (CTT) at 3 months and 9 months | baseline, 3-months, 9-months
  Colour Trails Tests (CTT) 1 and 2 assesses sustained attention and sequencing.
Change from baseline Block Design at 3 months and 9 months | baseline, 3-months, 9-months
  Block Design is a subtest that is administered as part of several of the Wechsler Intelligence tests, and it primarily measures visual-spatial and organizational processing abilities, as well as non-verbal problem-solving skills.
Change from baseline Semantic Verbal Fluency (Animals) at 3 months and 9 months | baseline, 3-months, 9-months
  Semantic Verbal Fluency (Animals) taps lexical knowledge and semantic memory organization.
Change from baseline fMRI scan at 3 months | baseline, 3-months
  Functional Magnetic Resonance Imaging (fMRI) will be employed to examine changes in functional connectivity. Images will be acquired on a 3T Siemens scanner using a standard Siemens whole head coil. All subjects will undergo the task-free fMRI scan after being instructed only to remain awake with their eyes closed. White Matter Diffiusion Tractography Imaging (DTI) will be utilized to identify anatomical connections between functionally correlated regions . The MRI Brain Scan is non-invasive and does not involve the use of Contrast; duration of each scan is approximately one hour.
Change from baseline Biomarkers: blood sample at 3 months and 9 months | baseline, 3-months, 9-months
  5 ml of blood will be collected using plasma tubes with indomethacin (15uM final conc) and BHT (20ul of 2mM) will be added prior to freezing (-80 Degree Celsius) to preserve the sample and prevent artifacts (at baseline, 3 months, 9 months).
  3 ml of blood will be collected using tubes with no coagulant (at baseline, 3 months and 9 months).
  5 ml of blood will be collected using Tempus Blood RNA tubes and will be stored in a refrigerator at approximately 4 Degree Celsius (at baseline and 9 months).
  Blood sample would be analysed for cytokine levels; chromosomal studies and terminal telomere restriction fragment length.
Change from baseline Biomarkers: urine sample at 9 months | baseline, 9-months
  15 ml sample of urine will be collected and frozen as quickly as possible. Urine sample would be analysed for oxidative biomarkers.
Change from baseline Biomarker - fecal sample at 3 months and 9 months | baseline,3 months, 9 months
  A fecal sample will also be collected in a tube with RNALater and microbeads. These can be kept at 40C till processing. Fecal sample would be analysed for bacteria.
Change from baseline Biomarker - saliva sample at 3 months and 9 months | baseline,3 months, 9 months
  Saliva will be collected in a test-tube by having participants continuously spit into a 50ml centrifuge tube for 5 minutes. Saliva sample would be analysed for salivary cortisol analysis, DNA extraction and sequencing for stress biomarkers (cytokines).

SECONDARY OUTCOMES:
Change from baseline Basic Health Screen at 3 months and 9 months | baseline, 3-months, 9-months
  the Blood pressure, Pulse rate, Height and Weight will be measured.
Change from baseline Activities of daily Living (ADL) at 3 months and 9 months | baseline, 3-months, 9-months
  Activities of daily Living (ADL) is a questionnaire to screen for functional assessment.
Change from baseline Instrumental Activities of Daily Living (IADL) at 3 months and 9 months | baseline, 3-months, 9-months
  Instrumental Activities of Daily Living (IADL) is a questionnaire to screen for functional assessment.
Change from baseline Geriatric Depression Scale (GDS) at 3 months and 9 months | baseline, 3-months, 9-months
  Psychological well-being will be assessed using the Geriatric Depression Scale. Subjects with high scores will not be enrolled into the study and will be informed of the scores and advised to see a doctor at a polyclinic or their family physician with a referral letter prepared for this purpose.
Change from baseline Geriatric Anxiety Inventory (GAI) at 3 months and 9 months | baseline, 3-months, 9-months
  Psychological well-being will be assessed using the Geriatric Anxiety Inventory (GAI). Subjects with high scores will not be enrolled into the study and will be informed of the scores and advised to see a doctor at a polyclinic or their family physician with a referral letter prepared for this purpose.

OTHER OUTCOMES:
Demographic questionnaire | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, Ph.D, Principal Investigator — National University of Singapore
Locations (1):
- Training and Research Academy, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Roberts RO, Geda YE, Knopman DS, Boeve BF, Christianson TJ, Pankratz VS, Kullo IJ, Tangalos EG, Ivnik RJ, Petersen RC. Association of C-reactive protein with mild cognitive impairment. Alzheimers Dement. 2009 Sep;5(5):398-405. doi: 10.1016/j.jalz.2009.01.025. PMID 19751919
- [Background] Moverare-Skrtic S, Johansson P, Mattsson N, Hansson O, Wallin A, Johansson JO, Zetterberg H, Blennow K, Svensson J. Leukocyte telomere length (LTL) is reduced in stable mild cognitive impairment but low LTL is not associated with conversion to Alzheimer's disease: a pilot study. Exp Gerontol. 2012 Feb;47(2):179-82. doi: 10.1016/j.exger.2011.12.005. Epub 2011 Dec 22. PMID 22210159
- [Background] Huang L, Jia J, Liu R. Decreased serum levels of the angiogenic factors VEGF and TGF-beta1 in Alzheimer's disease and amnestic mild cognitive impairment. Neurosci Lett. 2013 Aug 29;550:60-3. doi: 10.1016/j.neulet.2013.06.031. Epub 2013 Jul 1. PMID 23827227
- [Background] Gard T, Holzel BK, Lazar SW. The potential effects of meditation on age-related cognitive decline: a systematic review. Ann N Y Acad Sci. 2014 Jan;1307:89-103. doi: 10.1111/nyas.12348. PMID 24571182
- [Background] Rapgay L, Bystrisky A. Classical mindfulness: an introduction to its theory and practice for clinical application. Ann N Y Acad Sci. 2009 Aug;1172:148-62. doi: 10.1111/j.1749-6632.2009.04405.x. PMID 19735247
- [Background] Mcbee, L. (2008) Mindfulness-based elder care. New York: Springer.
- [Background] Wells RE, Yeh GY, Kerr CE, Wolkin J, Davis RB, Tan Y, Spaeth R, Wall RB, Walsh J, Kaptchuk TJ, Press D, Phillips RS, Kong J. Meditation's impact on default mode network and hippocampus in mild cognitive impairment: a pilot study. Neurosci Lett. 2013 Nov 27;556:15-9. doi: 10.1016/j.neulet.2013.10.001. Epub 2013 Oct 10. PMID 24120430
- [Background] Davidson RJ, Kabat-Zinn J, Schumacher J, Rosenkranz M, Muller D, Santorelli SF, Urbanowski F, Harrington A, Bonus K, Sheridan JF. Alterations in brain and immune function produced by mindfulness meditation. Psychosom Med. 2003 Jul-Aug;65(4):564-70. doi: 10.1097/01.psy.0000077505.67574.e3. PMID 12883106
- [Background] Feng L, Chong MS, Lim WS, Ng TP. The Modified Mini-Mental State Examination test: normative data for Singapore Chinese older adults and its performance in detecting early cognitive impairment. Singapore Med J. 2012 Jul;53(7):458-62. PMID 22815014
- [Background] Schmidt, M. (1996). Rey auditory verbal learning test: A handbook. Los Angeles: Western Psychological Services.
- [Background] Conway AR, Kane MJ, Bunting MF, Hambrick DZ, Wilhelm O, Engle RW. Working memory span tasks: A methodological review and user's guide. Psychon Bull Rev. 2005 Oct;12(5):769-86. doi: 10.3758/bf03196772. PMID 16523997
- [Background] Lee TM, Chan CC. Are trail making and color trails tests of equivalent constructs? J Clin Exp Neuropsychol. 2000 Aug;22(4):529-34. doi: 10.1076/1380-3395(200008)22:4;1-0;FT529. PMID 10923062
- [Background] Ardila, A., Ostrosky-Solís, F, & Bernal,B. (2006). Cognitive testing toward the future: The example of Semantic Verbal Fluency (ANIMALS), International Journal of Psychology, 41(5), 324-332
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Dusek JA, Otu HH, Wohlhueter AL, Bhasin M, Zerbini LF, Joseph MG, Benson H, Libermann TA. Genomic counter-stress changes induced by the relaxation response. PLoS One. 2008 Jul 2;3(7):e2576. doi: 10.1371/journal.pone.0002576. PMID 18596974